CLINICAL TRIAL: NCT02118155
Title: Connective Tissue Graft Associated or Not With Low Intensity Laser Therapy: A Randomized Clinical Trial
Brief Title: Low-intensity Laser Therapy in the Treatment of Gingival Recession
Acronym: LILT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, PhD, UPECLIN HC FM Botucatu Unesp
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0978412.5.0000.0077
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Connective tissue graft (CTG) (Sham Comparator): The gingival recession defects were treated by connective tissue graft surgical procedure and received the sham application os low-intensity laser therapy.
  Interventions: Procedure: Connective tissue graft
- Connective tissue graft plus laser (CTG+L) (Experimental): The gingival recession defects were treated by connective tissue graft associated with the application of a LILT protocol
  Interventions: Procedure: Connective tissue graft

INTERVENTIONS:
Procedure: Connective tissue graft — Periodontal surgical technique to treat gingival recessions

SUMMARY:
The purpose of this study was to evaluate the 6-month outcomes of applying low-intensity laser therapy associated with connective tissue grafts to treat gingival recession.

DETAILED DESCRIPTION:
This was a prospective, parallel and controlled clinical trial. The population evaluated in this study was selected at ICT - São José dos Campos, College of Dentistry.

The selected patients were randomly allocated (by a computer generated list) into:

Group CTG (n = 20) - patients who received connective tissue graft to treat gingival recession Group CTG+LILT (n = 20) - patients who received connective tissue graft associated with 8 applications of low-intensity laser therapy to treat gingival recession.

The surgeries, as well as all postoperative follow-up, were performed at the dental clinic of ICT- UNESP. Surgical areas were anesthetized (2% mepivacaine with 1:100,000 epinephrine). Two horizontal incisions were made at right angles to the adjacent interdental papillae, at the level of the CEJ, without interfering with the gingival margins of neighboring teeth. Two oblique vertical incisions were extended beyond the mucogingival junction, and a trapezoidal mucoperiosteal flap was raised up to the mucogingival junction. After this point, a split-thickness flap was extended apically, releasing the tension and favoring coronal positioning of the flap. The exposed root surface was gently scaled and planed to remove any possible irregularities. Afterward, a thin and small connective tissue graft was harvested from the palate using a scalpel with parallel blades (1.0 mm away from each other). The graft was sutured# using single sutures in the papillae, over the root surface, in such a way that covered the CEJ and the recession. Then, the flap was coronally positioned and sutured to completely cover the graft The patients allocated for the test group received the following protocol for laser application: Five (5) points of irradiation were performed, as depicted in Figure 1. The irradiation was performed with a GaAlAs** diode laser that continuously emitted a wavelength of 660 nm. 30 mW was used for 20 seconds, and the total applied energy density (fluence) was 15 J/cm2 (3 J/cm2 per point and an application time of 4 seconds per point)

Clinical parameters were assessed at baseline and 3 and 6 months post-operatively.

Statistical Analysis The null hypothesis considered in the study was the absence of difference in the clinical parameters between the different groups. For data analysis, the statistical program was used (Sigmaplot). The demographic and clinical data were compared between the groups using Student's t-test. The data were first analyzed for homogeneity using the Shapiro-Wilk test, which indicated non-normal distribution. . Those presenting Shapiro-Wilk p values < 0.05 were analyzed using a Friedman test (for intragroup comparisons) and Mann-Whitney tests (for intergroup comparisons). Patients' esthetics and discomfort measures using VAS were analyzed by T-tests. The frequency of sites that were scored as very good or excellent in each group by QCE analysis, the frequency of complete root coverage, BOP, and the presence or absence of plaque at the site were compared using χ2 tests. Intergroup RES comparisons were performed with a T-test. A significance level of 0.05 was adopted.

ELIGIBILITY:
Inclusion Criteria:

1. presenting Miller class I or II gingival recession in the maxillary canines or premolars;
2. visible cemento-enamel junction (CEJ) in the teeth included in the study and pulp vitality;
3. patients presenting no signs of active periodontal disease and full-mouth plaque and bleeding score ≤ 20%;
4. patients older than 18 years old;
5. probing depth ˂ 3 mm in the included teeth; 6) patients who agreed to participate and signed an informed consent form

Exclusion Criteria:

1. patients with systemic problems (cardiovascular, blood dyscrasias, immunodeficiency, and diabetes, among others) that will contraindicate the surgical procedure
2. patients taking medications known to interfere with the wound healing process or that contraindicate the surgical procedure
3. smokers or pregnant women
4. patients who underwent periodontal surgery in the area of interest; and 5) patients with orthodontic therapy in progress.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Percentage of root coverage | 6 months

SECONDARY OUTCOMES:
Esthetic | 6 months
  Two esthetic evaluations were performed: 1 professional and 1 patient-centered. The professional esthetic evaluation was made using the photographs of the baseline and 6 months after surgery set in a before-and-after panel. The professional evaluation was conducted using the root coverage esthetic score (RES).
  Esthetic outcomes were also evaluated from the patient's point of view. Using a hand mirror, the patients viewed the gingival recession before and after 6 months and were asked to rate the esthetics of the tooth included in the study on a VAS scale.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie B Fernandes-Dias, DDS, Ms, Study Chair — UPECLIN HC FM Botucatu Unesp; Maria Aparecida N Jardini, PhD, Study Chair — UPECLIN HC FM Botucatu Unesp
Locations (1):
- UNESP - ICT Odontologia São José dos Campos, São José dos Campos, São Paulo, Brazil

REFERENCES:
- [Background] Ozturan S, Durukan SA, Ozcelik O, Seydaoglu G, Haytac MC. Coronally advanced flap adjunct with low intensity laser therapy: a randomized controlled clinical pilot study. J Clin Periodontol. 2011 Nov;38(11):1055-62. doi: 10.1111/j.1600-051X.2011.01774.x. Epub 2011 Sep 15. PMID 22092477
- [Derived] Santamaria MP, Fernandes-Dias SB, Araujo CF, Lucas da Silva Neves F, Mathias IF, Rebelato Bechara Andere NM, Neves Jardini MA. 2-Year Assessment of Tissue Biostimulation With Low-Level Laser on the Outcomes of Connective Tissue Graft in the Treatment of Single Gingival Recession: A Randomized Clinical Trial. J Periodontol. 2017 Apr;88(4):320-328. doi: 10.1902/jop.2016.160391. Epub 2016 Nov 11. PMID 27834120
- [Derived] Fernandes-Dias SB, de Marco AC, Santamaria M Jr, Kerbauy WD, Jardini MA, Santamaria MP. Connective tissue graft associated or not with low laser therapy to treat gingival recession: randomized clinical trial. J Clin Periodontol. 2015 Jan;42(1):54-61. doi: 10.1111/jcpe.12328. Epub 2014 Dec 17. PMID 25363203